CLINICAL TRIAL: NCT05091931
Title: A Prospective Observational Cohort Study Comparing the Effects of Guidance® UTI vs. Culture-based Testing Methods on Antibiotic Prescribing Practices in an Outpatient Setting
Brief Title: Diagnosis, Antibiotic Prescribing Practices and Outcomes of cUTI in an Outpatient Setting
Status: Completed | Type: Observational
Sponsor: Pathnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-UTI-PMAS
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Urinary Tract Infections
Keywords: Recurrent UTI; Complicated Urinary Tract Infection; C Difficile; Adverse Drug Event
MeSH Terms: conditions — Urinary Tract Infections; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Data or specimens collected in this research study might be used for future research or distributed to another investigator for future research without your consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Guidance® UTI pathway (standard lab workflow): Guidance® UTI pathway with antibiotic sensitivity and microbial testing results available to ordering provider within 48 hours of lab receipt. Includes confirmation by the clinical lead that the ordering provider has acted upon results as soon as they are made available. The lab will follow current workflows in terms of result reporting. Treatment based on local standard clinical antibiotic selection with or without empiric therapy.
- Guidance® UTI pathway (modified lab workflow): Guidance® UTI pathway with antibiotic sensitivity and microbial testing results reporting to a clinical lead specialist at the urology office within 14 hours of lab receipt. Includes confirmation by the clinical lead that the ordering provider has acted upon results as soon as they are made available. Treatment based on local standard clinical antibiotic selection with or without empiric therapy.
- Traditional clinical pathway: Local standard clinical practice pattern for UTI testing (e.g., urine analysis, urine culture and sensitivities or molecular testing as available). Treatment based on local standard clinical antibiotic selection with or without empiric therapy

SUMMARY:
This prospective, multicenter, comparative cohort observational study is to determine if Guidance® UTI pathway compared to traditional diagnostic pathways reduces the rates of empiric antibiotic therapy, adverse events, and improves therapeutic accuracy of treatment

DETAILED DESCRIPTION:
We propose to conduct a multicenter, comparative cohort observational study to determine whether the use of Guidance® UTI Clinical Pathway compared with current traditional pathways for urine testing reduces the rates of empiric antibiotic therapy and improves therapeutic accuracy of treatment. Comparative outpatient Urology and urogynecology office cohorts will be allocated at an uneven 2:1 allocation ratio. Regardless of arm assignment, all outpatient offices have the option to order ANY diagnostic test for suspected UTI, this includes urine cultures and/or other molecular testing methods including Guidance® UTI. If a provider in the Guidance Clinical Pathway arm decides to order urine cultures instead of using the Guidance® UTI Clinical Pathway, those results will also be reported to the site lead, though TAT may take up to 72 hours to result per standard culture protocols. We will be observing the practice's implementation of the Clinical Pathway and reporting infrastructure to provide rapid, centralized reporting to the ordering provider, allowing for efficient treatment. Guidance® UTI is currently widely available, and all participating outpatient offices (regardless of arm) will have the option to order this test.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide verbal informed consent
* Male and Female Subjects > 18 years of age may participate with no predetermined quotas or ratios for gender participation (Group 2).
* Male and Female Subjects > 18 and older may participate with no predetermined quotas or ratios for gender participation (Group 1).
* A history of complicated UTI (cUTI)**
* Must present at the time of enrollment with clinically suspected active UTI (any LUTS)
* Management requires microbial identification and sensitivities of urine

  **Definition of cUTI- A UTI is considered complicated when the individual has one or more risk factors that predispose to higher treatment failure and poor outcomes.6 These poor outcomes include persistence of UTI, increasing severity, or occurrence of complications such as urosepsis, recurrence, and perinephric abscess. Although the definition of cUTI may vary among current medical bodies and organizations, for this study, we define examples of cUTIs to include:
* UTIs in the elderly population due to increased chances of comorbidities and immune compromised state,
* Recurrent UTIs2, which is defined as the occurrence of ⩾2 symptomatic episodes within 6 months or ⩾3 symptomatic episodes within 12 months
* UTI in patients with anatomic or functional pathology affecting the urinary tract, such as an obstruction, hydronephrosis, renal tract calculi, or colovesical fistula
* UTIs occurring due to an immune compromised state, such as steroid use, post chemotherapy, diabetes, and HIV, and transplant recipients
* UTIs caused by atypical microorganisms or multi-drug resistant microorganisms. Typical UTI-causing microorganisms include E. coli, P. aeruginosa, several species within the Enterobacteriaceae family (Proteus and Klebsiella), and a few Gram- positive bacteria, such as Staphylococcus saprophyticus and Enterococcus faecalis, as well as fungi, such as Candida sp.7,5
* UTI in male: UTIs occurring despite the presence of anatomical protective measures as part of the male urinary tract anatomy are by definition cUTI,
* UTI in patients with history of radiotherapy to the abdomen or pelvis,
* UTIs occurring after instrumentation, nephrostomy tubes, ureteric stents, suprapubic tubes, or Foley catheters
* UTI in patients with the history of recurrent UTI,
* UTIs in patients with impaired renal function,
* UTIs following prostatectomies or radiotherapy

Exclusion Criteria:

* Patients with history of chronic pelvic pain syndrome/interstitial cystitis (Excluded in GROUP 2 only)
* Patients that are receiving radiation therapy in the pelvic region
* Patients with history of unstable, untreated, or are failing treatment for overactive bladder (either neurogenic or non-neurogenic)
* Patients with history of bladder malignancy in the past 3 years
* Patients that have been treated with chemotherapy in the past 3 years
* Inability to independently provide symptom data
* Patient must have email access if they choose to complete surveys online.
* Pregnancy
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals >18 years requiring evaluation for suspected urinary tract infection in the urology or urogynecology practice.
Sampling Method: Non-Probability Sample
Enrollment: 3308 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
The percentage of outpatients seen for suspected UTI started on empiric treatment | 30 days
  The percentage of outpatients seen for suspected UTI started on empiric treatment
Rate of Adverse Events through 30 days | 30 days
  The incidence rate of the adverse events (listed below) 30 days following index visit.
  * Allergic reactions to antibiotic therapy
  * Nausea/vomiting, headache, skin rash, anaphylaxis/hypersensitivity reaction
  * yeast infection (Vaginitis/vulvovaginal candidiasis)
  * Acute renal failure
  * tendinopathy (including tendon rupture)
  * C. difficile infection
  * ED Visit/Urgent care (UTI)
  * Hospitalization (UTI)
  * Sepsis
  * Recurrent UTI (rUTI) - The proportion of subjects reporting recurrence of symptomatic UTI and receive antimicrobial treatment (re-prescription). All subjects having reported initial resolution of their UTI symptoms by day 14 will be assessed for this outcome.

SECONDARY OUTCOMES:
Resolution of the Initial UTI Symptoms by Day 14 | 14 Days
  Patients will be asked about UTI symptoms on days 1- 14 after index visit. Patients showing improvement in overall symptom score over 14 days versus baseline score. Subjects with persistent UTI symptoms or having received further antimicrobials because of UTI symptoms will be considered to have not met the outcome, whereas those without persistent UTI symptoms and not having received further antimicrobials will be considered to have met the outcome.
Resolution of Symptoms | 30 days
  Complete Resolution of symptoms by day 30
Antibiotics Concordance with Sensitivity Results | 30 days
  Percentage of prescribed antibiotics that are concordant with sensitivity results
Biomarkers | 30 days
  Number of samples containing biomarker concentration above specific thresholds; unique to each biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Baunoch, PhD, Principal Investigator — Clinical Trials
Locations (2):
- United States (2):
  - First Urology, Louisville, Kentucky
  - Comprehensive Urology, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No